CLINICAL TRIAL: NCT06611488
Title: Effect of Sleep Disturbances on Postural Control in the Elderly Population
Brief Title: Sleep Disturbances on Postural Control in the Elderly Population
Status: Completed | Type: Observational
Sponsor: Shaimaa Mohamed Ahmed Elsayeh (Other)
Collaborators: Majmaah University (Other)
Responsible Party: Sponsor-Investigator, Shaimaa Mohamed Ahmed Elsayeh, Assistant Professor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: MUREC-March. I 7/COM -202 I /2
Record Dates: First submitted 2024-09-10; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Sleep Quality; Postural Stability
Keywords: Sleep disturbances; Postural control; Elderly population
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal sleepiness group: Participants with normal daytime sleepiness
  Interventions: Other: No Intervention: Observational Cohort
- Excessive daytime sleepiness group: Participants with excessive daytime sleepiness group
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention as the study is bservational Cohort

SUMMARY:
The sleep disorders are common among older adults and comprises of wide spectrum of the sleep related issues like poor sleep quality, sleep deprivation and excessive day time sleepiness.

DETAILED DESCRIPTION:
Earlier studies were carried to determine the effect of sleep deprivation on the postural control parameters. The effect of poor sleep quality and excessive daytime sleepiness on the postural control were not widely studied. Aim : To determine the effect of the sleep quality and excessive daytime sleepiness on the postural stability during quiet standing and whether this influence vary based on the availability of the visual feedback.

ELIGIBILITY:
Inclusion Criteria:

* Be able to stand unsupported with eyes opened and eyes closed for 30 seconds.

Exclusion Criteria:

* Elderly with uncorrected visual impairment, Underwent bilateral hip replacement.
* Participants using drugs which affect control.
* Participants with previous history of conditions which affect postural control.

Min Age: 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly participant with age 67 years and more
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Postural stability using STABLE platform | "Immediately after enrollment"
  The Postural stability of the participants was assessed using STABLE by Motek medical that made in Netherlands. During each trial, participants were made to stand quietly for 30 seconds on the platform of STABLE with open eyes first and after that with closed eyes "Individuals should initially complete two sessions of test with open eyes, then followed with closed eyes". And after that comparison of postural stability between both normal sleepiness and excessive daytime sleepiness groups.

OTHER OUTCOMES:
Sleep parameters using the Arabic version of Pittsburgh Sleep Quality Index | "Immediately after enrollment"
  The Arabic version of Pittsburgh Sleep Quality Index (PSQI), it's a self-administered validated questionnaire to ass the quality of sleep over previous weeks. The PSQI is comprehensive and consists of 19 items combined into seven subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications and daytime dysfunction. The scores of each component range from 0 to 3 and global or total PSQI score is calculated by summing all the scores of all seven components yielding a maximum possible score of 21. The higher scores reflecting poor sleep quality. In the current study, the cut-off score of more than 5 to categorize as poor sleep quality. It also will be used to align the participants to either normal sleepiness group or excessive day time sleepiness group.
Day time sleepiness using The Arabic version of Epworth Sleepiness Scale. | "Immediately after enrollment"
  The Arabic version of Epworth Sleepiness Scale (ESS) was administered to determine the daytime sleepiness The ESS necessitates the user to report the chance of dozing as per four-point scale [0 indicates no chance of dosing, 1 indicates slight chance of dozing, 2 indicates moderate chance of dozing, 3 indicates high chance of dozing] in eight given situations. The scores of the ESS range from 0 to 24, higher scores demonstrating excessive daytime sleepiness. In the current study, the cut-off score of more than 10 to categorize as excessive daytime sleepiness. It will be used to align the participants to either normal sleepiness group or excessive day time sleepiness group.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrhman Y Alqahtani, Master degree, Principal Investigator — The Majmaah University; Zeinab A Ali, PhD, Study Director — Cairo University; Shaimaa M Elsayeh, PhD, Study Director — Cairo University
Locations (1):
- The Majmaah University, Al Majmaah, Riyadh/ Saudi Arabia, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melzer I, Benjuya N, Kaplanski J. Age-related changes of postural control: effect of cognitive tasks. Gerontology. 2001 Jul-Aug;47(4):189-94. doi: 10.1159/000052797. PMID 11408723